CLINICAL TRIAL: NCT07340398
Title: Neoadjuvant Trastuzumab-rezetecan Plus Pertuzumab or Nab-Paclitaxel, Carboplatin, Trastuzumab, and Pyrotinib After Suboptimal Response to Neoadjuvant Dual HER2-Targeted Therapy Combined With Chemotherapy in HER2-Positive Early Breast Cancer: A Response-Guided Phase II Study (TAYLOR)
Brief Title: Neoadjuvant Trastuzumab-rezetecan Plus Pertuzumab or Nab-Paclitaxel, Carboplatin, Trastuzumab, and Pyrotinib After Suboptimal Response to Neoadjuvant Dual HER2-Targeted Therapy Combined With Chemotherapy in HER2-Positive Early Breast Cancer
Acronym: TAYLOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1587
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: HER2-positive Early Breast Cancer
MeSH Terms: interventions — Taxes; Carboplatin; Trastuzumab; pertuzumab; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nab-PCbHPy (Experimental)
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pyrotinib
- SHR-A1811+P (Experimental)
  Interventions: Drug: Pertuzumab; Drug: SHR-A1811

INTERVENTIONS:
Drug: Nab paclitaxel — Nab paclitaxel
  Arms: nab-PCbHPy
Drug: Carboplatin — carboplatin
  Arms: nab-PCbHPy
Drug: Trastuzumab — trastuzumab
  Arms: nab-PCbHPy
Drug: Pertuzumab — pertuzumab
  Arms: SHR-A1811+P
Drug: SHR-A1811 — a HER2-targeted antibody-drug conjugate (ADC)
  Other Names: Trastuzumab-rezetecan
  Arms: SHR-A1811+P
Drug: Pyrotinib — Pyrotinib: an oral irreversible pan-HER tyrosine kinase inhibitor (TKI).
  Arms: nab-PCbHPy

SUMMARY:
This prospective, response-guided phase II study investigates individualized neoadjuvant treatment strategies for patients with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer. After receiving neoadjuvant dual-HER2-targeted therapy with chemotherapy, patients are evaluated for their treatment response. Those achieving an adequate response continue the therapy, whereas patients with a suboptimal response transition to an intensified investigational regimen incorporating novel targeted agents. This adaptive approach aims to optimize pathologic response, minimize unnecessary toxicity, and explore more effective treatment options for individuals with insufficient benefit from conventional neoadjuvant therapy.

DETAILED DESCRIPTION:
This is a prospective, response-guided, phase II study designed to evaluate individualized neoadjuvant treatment strategies in patients with HER2-positive early breast cancer. The study incorporates an adaptive treatment algorithm based on early response assessment to an initial neoadjuvant dual HER2-targeted therapy combined with chemotherapy, with the aim of optimizing therapeutic efficacy while minimizing unnecessary treatment-related toxicity.

All eligible patients initially receive neoadjuvant dual HER2-targeted therapy combined with chemotherapy according to the study protocol. Following completion of a predefined initial treatment phase, tumor response is systematically assessed using standardized clinical and radiologic criteria.

Patients who achieve an adequate response continue the same neoadjuvant treatment to complete the planned course of therapy. In contrast, patients demonstrating a suboptimal response are assigned to an intensified investigational neoadjuvant strategy. The escalation regimens include either trastuzumab-rezetecan in combination with pertuzumab or a pyrotinib-based multi-agent regimen incorporating chemotherapy and HER2-directed therapy. Treatment selection and administration follow protocol-specified criteria and schedules.

The response-guided escalation strategy is intended to address the unmet clinical need of patients who derive insufficient benefit from standard neoadjuvant dual HER2-targeted therapy combined with chemotherapy. By selectively intensifying treatment only in patients with suboptimal response, this study seeks to enhance pathologic response rates while avoiding overtreatment in patients who respond adequately to initial therapy.

Primary and secondary objectives focus on evaluating pathologic response outcomes, safety and tolerability of the adaptive treatment strategies, and feasibility of response-guided treatment modification in the neoadjuvant setting. Exploratory analyses will assess potential biomarkers associated with treatment response and resistance, providing insights to inform future personalized neoadjuvant treatment approaches in HER2-positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
3. Primary tumor size >1 cm.
4. Histologically confirmed invasive breast cancer, clinically staged as:

   * Stage I (T1cN0M0)
   * Stage II (T1cN1M0, T2N0-1M0 or T3N0M0)
   * Stage III (T2N2-3M0, T3N1-3M0, or T4N0-3M0)
5. HER2-positive status: IHC 3+ or IHC 2+ with positive ISH.
6. Adequate major organ function:

   1. Hematology (no transfusion or hematopoietic growth factors, e.g., G-CSF, within 14 days):

      * Hemoglobin ≥100 g/L
      * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L
      * Platelet count ≥100 × 10⁹/L
   2. Biochemistry:

      * Total bilirubin ≤1.5 × ULN
      * ALT and AST ≤1.5 × ULN; ALP ≤2.5 × ULN
      * BUN and creatinine ≤1.5 × ULN
   3. Cardiac function: LVEF ≥55% by echocardiography
7. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment and agree to use effective contraception during the study and for 8 weeks after the last dose.
8. Voluntary written informed consent and willingness to comply with study procedures and follow-up.

Exclusion Criteria:

1. Prior anti-tumor therapy for breast cancer, including chemotherapy, radiotherapy, targeted therapy, or endocrine therapy.
2. Concurrent administration of any other anti-tumor treatment.
3. Bilateral breast cancer, inflammatory breast cancer, or occult breast cancer.
4. Breast cancer not confirmed histologically.
5. History of other malignancy within the past 5 years, except successfully treated cervical carcinoma in situ.
6. Severe dysfunction of major organs (heart, liver, kidney).
7. Conditions affecting oral drug administration or absorption, e.g., inability to swallow, chronic diarrhea, or intestinal obstruction.
8. Participation in another investigational drug trial within 4 weeks prior to enrollment.
9. Known hypersensitivity to study drug components; history of immunodeficiency (HIV positive, active HCV, active hepatitis B, other congenital/acquired immunodeficiency) or prior organ transplantation.
10. History of clinically significant cardiac disease, including:

    1. Arrhythmia requiring medication
    2. Myocardial infarction
    3. Heart failure
    4. Other cardiac conditions deemed unsuitable for study participation by the investigator
11. Pregnant or breastfeeding women, or women of childbearing potential who test positive at baseline or are unwilling to use effective contraception throughout the study.
12. Any condition that, in the investigator's judgment, poses serious risk to patient safety or may interfere with study completion (e.g., uncontrolled severe hypertension, uncontrolled diabetes, active infection).
13. History of neurological or psychiatric disorders (e.g., epilepsy or dementia) or any other condition the investigator considers incompatible with study participation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Pathological Complete Response (tpCR) Rate: ypT0/Tis, ypN0 | 18 weeks
  The tpCR rate is defined as the proportion of participants with no residual invasive cancer cells in both the breast primary tumor site (residual in situ cancer cells are permitted) and all sampled axillary lymph nodes.

SECONDARY OUTCOMES:
Breast Pathological Complete Response (bpCR) Rate: ypT0/Tis | 18 weeks
  The bpCR rate is defined as the proportion of participants with no residual invasive cancer cells in the breast primary tumor site (residual in situ cancer cells are permitted).
Objective Response Rate (ORR) | 18 weeks
  ORR is defined as the proportion of participants with a complete or partial response.
Event-Free Survival (EFS) | Approximately five years
  EFS is defined as the time from randomization to any of the following events: precludes surgery, local or distant recurrence, second primary malignancy, or death due to any cause.
Adverse Event (AE) | Approximately three years
  An AE is defined as any untoward medical occurrence in a study participant administered a medicinal product, temporally associated with study intervention, without presumption of causality.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China